CLINICAL TRIAL: NCT01063725
Title: A Multi-center, Randomized, Placebo-controlled Double Blind Clinical Study Assessing the Efficacy and Safety of Femarelle® in Menopausal Women With Vasomotor Syndrome
Brief Title: A Double-Blind Study to Evaluate the Effect of Femarelle® on Menopausal on Vasomotor Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Se-cure Pharmaceuticals Ltd. (Industry)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FS1
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2010-02

CONDITIONS: Menopause; Hot Flashes
Keywords: menopause; hot flashes; vasomotor symptoms; femarelle; soy extract; SERM
MeSH Terms: conditions — Hot Flashes | interventions — DT56a; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femarelle (Experimental): Women will receive Femarelle twice daily for 12 weeks
  Interventions: Dietary Supplement: Femarelle
- Placebo (Placebo Comparator): Women will take placebo capsules twice daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Femarelle — A soy based food supplement containing 322 mg of soy extract and 108 mg of flaxseed, to be taken twice daily
  Other Names: Tofupill
  Arms: Femarelle
Other: Placebo — Capsules containing 430 mg of microcrystalline cellulose, as a placebo, to be taken twice daily
  Other Names: Avicel
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effects of Femarelle ( a plan-derived SERM) on hot flushes and quality of life in menopausal women. Our hypotheses are that compared to placebo, Femarelle reduces the daily number of hot flushes and their severity and also improves the quality of life as measured by validated dairies and questionnaires.

DETAILED DESCRIPTION:
Symptomatic menopausal women will be divided to treatment with Femarelle or placebo for 12 weeks after two weeks of baseline record. Hot flashes daily diary will be recorded daily and a quality of life questionnaire will be filled at the beginning and at completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. postmenopausal women, i.e 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/
2. More than 7 hot flushes per day or over 50 per week at baseline.
3. Women should have documentation of a negative screening mammogram (obtained at screening or within 1 year of study enrolment.
4. Normal pelvic and breast exams by investigator prior to enrolment.
5. All subjects who have a uterus should have endometrial thickness of less than 5mm in vaginal sonogram exam at randomization.
6. Informed consent to participate in the study.

Exclusion Criteria:

1. Use of any medication or supplements for menopausal symptoms, such as estrogen/progestin containing drug products, Isoflavons, phytoestrogens and SERM within a minimum of 8 weeks prior to pre-study screening period.
2. Use of SSRIs, St. John's Wort, within a minimum of 8 weeks prior to pre-study screening period.
3. Any clinically unstable or uncontrolled renal, hepatic, endocrine, respiratory, hematological, neurological, cardiovascular or cerebrovascular disease that would put the subject at safety risk or mask measure of efficacy
4. Evidence or history of vascular disease (such as ischemic heart disease), Cerebrovascular accident (such as stroke or transient ischemic attack) or deep vein thrombosis (blood clots), or thromboembolic disorders.
5. Personal history of breast cancer
6. Abnormal clinically relevant vaginal bleeding
7. Any clinically relevant (opinion of investigator) abnormal finding during physical, gynecological and breast examination at screening
8. Abnormal, clinically significant results of mammography
9. Malignancy with the exception of BCC of the skin
10. Known hypersensitivity to gluten, soybeans, soy protein, estrogens and/or progestins
11. History of severe recurrent depression, or severe psychiatric disturbance. Untreated or uncontrolled high blood pressure (hypertension)
12. Participation in a clinical trial within 30 days prior to screening Known substance abuse (alcohol or drug)
13. Unable to comply with study protocol

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 4 in the average Number of Hot Flashes per day | 4 weeks
Change from Baseline to Week 4 in the average daily Severity Score of hot flashes | 4 weeks
Change from Baseline to Week 12 in the average Number of Hot Flashes per day (averaged over the week) | 12 weeks
Change from Baseline to Week 12 in the average daily Severity Score of hot flashes | 12 weeks

SECONDARY OUTCOMES:
Change in average Number of Hot Flashes per day from Baseline to Week 4 and Week 12 | 12 weeks
No serious adverse event in either groups from Week 0 (Baseline) to Week 12. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bari Kaplan, Prof., Principal Investigator — Clalit Health Services
Locations (5):
- Israel (5):
  - Women's Health Center, Afula
  - Women's Health Clinic, Ashdod
  - Women's Health Clinic, Bet Shemesh
  - Women's Health Clinic, Bnei Brak
  - Women's Health Clinic, Rehovot